CLINICAL TRIAL: NCT03367039
Title: Clinical and Radiographic Analysis of ProDisc-C Vivo to Treat Degenerative Disc Disease: A 7-year Follow-up, Multi-center, Prospective, Randomized, Controlled Clinical Trial.
Brief Title: A Multi-center Prospective Randomized Controlled Study on Clinical and Radiographic Analysis of ProDisc-C Vivo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Zhenqi, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prodisc-C vivo
Record Dates: First submitted 2017-11-29; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Disk Degeneration; Cervical Disc Disease
Keywords: ProDisc-C vivo; ACDF; Cervical degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: 648 DDD patients (age from 20 to 70) from several hospitals matching the inclusion criteria will be randomly assigned to two groups (324 patients in each group). One group will be treated with ProDisc-C vivo disc replacement. The other groups will be treated with ACDF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProDisc-C vivo (Experimental): This group of patients will be treated with ProDisc-C vivo disc replacement (single segment).
  Interventions: Procedure: ProDisc-C vivo
- Anterior cervical discectomy fusion (Active Comparator): This group of patients will be treated with anterior cervical discectomy fusion (ACDF) procedure (single segment).
  Interventions: Procedure: Anterior cervical discectomy fusion

INTERVENTIONS:
Procedure: ProDisc-C vivo — Total Disc Replacement using ProDisc-C vivo.
  Arms: ProDisc-C vivo
Procedure: Anterior cervical discectomy fusion — Anterior Cervical Discectomy and Fusion
  Arms: Anterior cervical discectomy fusion

SUMMARY:
The object of this study is to assess the long-term safety and efficacy of cervical disc replacement with the ProDisc-C vivo Cervical Disc in a prospective, randomized, multi-center trial with 7 years of follow-up.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter trial at 7 years of follow-up comparing ProDisc-C vivo artificial cervical disc replacement and ACDF (Anterior cervical discectomy fusion) to treat degenerative disc disease (DDD). 648 DDD patients (age from 20 to 70) from several hospitals matching the inclusion criteria will be randomly assigned to two groups (324 patients in each group). One group will be treated with ProDisc-C vivo disc replacement. The other group will be treated with ACDF. The clinical outcomes and radiographic measurements will be compared between two groups at 1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Single-level cervical disc disease.
* At least one additional confirmatory neuroradiographic study, such as MRI or CT- enhanced myelography that showed findings consistent with clinical findings and complaints.

Exclusion Criteria:

* Patients have cervical spinal conditions other than single-level symptomatic degenerative disc disease or evidence of instability.
* Symptomatic disc disease at level C2 -3 or C7-T1.
* A history of discitis.
* A medical condition that required medication,such as steroids or nonsteroidal antiinflammatory medications that could interfere with fusion.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change of overall success rate | The overall success will be assessed at each time point (1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments).
  A patient's outcome was considered an overall success if all of the following conditions were met: 1) postoperative (Neck Disability Index) NDI score improvement of at least a 15-point increase from preoperative score; 2) maintenance or improvement in neurological status; 3) disc height success; 4) no serious adverse event classified as implant associated or implant/surgical procedure associated; and 5) no additional surgical procedure classified as a "failure".

SECONDARY OUTCOMES:
Change of sagittal angular motion | The radiographic outcomes will be obtained at each study point (before surgery,1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments).
  Neutral anteroposterior and lateral radiographs and dynamic flexion-extension lateral radiographs will be measured.
Change of neck disability index scores | The NDI scores will be obtained at each study point (before surgery,1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments).
  The neck disability index(NDI) questionnaire measures the level of pain and disability associated with various activities. The NDI is a 10-item, 50-point index that assesses different aspects of daily functioning in patients with neck pain. Each item is scored 0 to 5. The NDI score is a sum of the scores of the10-item. Clinical effects will be evaluated based on scores of the NDI. Higher values represent a better outcome.
Change of Arm and Neck pain intensity | Neck and arm pain scores will be measured at each study point (before surgery,1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments).
  Neck and arm pain scores will be measured using a visual analogue scale (VAS) from "0' (no sensation) to '100"(the most intense pain imaginable) where 30 means "pain threshold".

CONTACTS AND LOCATIONS:
Overall Officials: Zhenqi Zhu, Master, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sasso RC, Anderson PA, Riew KD, Heller JG. Results of cervical arthroplasty compared with anterior discectomy and fusion: four-year clinical outcomes in a prospective, randomized controlled trial. J Bone Joint Surg Am. 2011 Sep 21;93(18):1684-92. doi: 10.2106/JBJS.J.00476. PMID 21938372
- [Background] Steinmetz MP, Patel R, Traynelis V, Resnick DK, Anderson PA. Cervical disc arthroplasty compared with fusion in a workers' compensation population. Neurosurgery. 2008 Oct;63(4):741-7; discussion 747. doi: 10.1227/01.NEU.0000325495.79104.DB. PMID 18981885
- [Background] Mummaneni PV, Burkus JK, Haid RW, Traynelis VC, Zdeblick TA. Clinical and radiographic analysis of cervical disc arthroplasty compared with allograft fusion: a randomized controlled clinical trial. J Neurosurg Spine. 2007 Mar;6(3):198-209. doi: 10.3171/spi.2007.6.3.198. PMID 17355018